CLINICAL TRIAL: NCT06746636
Title: Comparison Between Four Weaning Methods from High-velocity Nasal Insufflation Device in Acute Hypoxemic Respiratory Failure
Acronym: HVNI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Hsanen, Lecturer of chest diseases and tuberculosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: weaning from HVNI
Record Dates: First submitted 2024-12-10; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure with Hypoxia
Keywords: HVNI; HFNC; HFNO; weaning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Flow reduction (Experimental): the flow will gradually be reduced by 10 L/ min/h. When it reaches 20 L/min, FiO2 reduction will then begin at 0.1 /h until it reaches 0.3.
  Interventions: Device: High velocity nasal insufflation
- Oxygen reduction (Experimental): FiO2 will gradually be reduced by 0.1 /h until it reaches 0.3. At this point, the flow will be reduced by 10 L/min/h until it reaches 20 L/min.
  Interventions: Device: High velocity nasal insufflation
- Sudden reduction (Experimental): HVNI will be abruptly discontinued after fulfilling weaning criteria provided that flow and Fio2 are less than 40 L\min and 40%
  Interventions: Device: High velocity nasal insufflation
- Flow and oxygen reduction (Experimental): both flow and FiO2 will be gradually reduced simultaneously at a rate of 10 L/min and 0.1 /h, respectively, until they reach 20 L/min for flow and 0.3 for FiO2
  Interventions: Device: High velocity nasal insufflation

INTERVENTIONS:
Device: High velocity nasal insufflation — • HVNI was supplied using a Vapotherm Precision Flow [Precision Flow Plus, Vapotherm, INC. U.S.A. device].

SUMMARY:
High-flow nasal oxygen therapy (HFNO) is an innovative high-flow system that allows for delivering up to 60 liters/ min of heated and fully humidified gas with a fraction of inspired oxygen (FIO2) ranging between 21% and 100% . High-flow nasal oxygen therapy has become an increasingly popular choice of therapy due to the potential complications of invasive ventilation and the frequent uncomfortable or life-threatening adverse effects that are produced in non-invasive ventilation (NIV) . The HFNO allows the modification of only two variables: the percentage of oxygen being delivered and the rate of gas flow . Numerous well-designed studies have been conducted into the use of the HFNC in the treatment of critically ill patients, and HFNC is now widely used in the treatment of patients with various diagnoses including acute hypoxemic respiratory failure or acute respiratory distress syndrome (ARDS) , and is used in post-extubation treatment, post-cardiothoracic surgery respiratory distress , and respiratory compromise induced by heart failure .

High-velocity nasal insufflation (HVNI) is a form of HFNC that utilizes a small bore nasal cannula to generate higher velocities of gas delivery than its counterparts using large bore HFNC. HVNI can accomplish a complete purge of extrathoracic dead space and may be able to provide ventilatory support in patients with acute hypercapnic respiratory failure in addition to oxygenation support.

This study is necessary because, even though studies were being conducted to determine both the optimal technique for HFNO delivery and the clinical setting in which it is most useful, the best strategy for weaning from HVNI remains unknown. It has also not been established at what point a patient should be considered stable enough to attempt for withdrawing the HVNI

DETAILED DESCRIPTION:
High-flow nasal oxygen therapy (HFNO) is an innovative high-flow system that allows for delivering up to 60 liters/ min of heated and fully humidified gas with a fraction of inspired oxygen (FIO2) ranging between 21% and 100% . High-flow nasal oxygen therapy has become an increasingly popular choice of therapy due to the potential complications of invasive ventilation and the frequent uncomfortable or life-threatening adverse effects that are produced in non-invasive ventilation (NIV) . The HFNO allows the modification of only two variables: the percentage of oxygen being delivered and the rate of gas flow . Numerous well-designed studies have been conducted into the use of the HFNC in the treatment of critically ill patients, and HFNC is now widely used in the treatment of patients with various diagnoses including acute hypoxemic respiratory failure or acute respiratory distress syndrome (ARDS) , and is used in post-extubation treatment , post-cardiothoracic surgery respiratory distress , and respiratory compromise induced by heart failure.

High-velocity nasal insufflation (HVNI) is a form of HFNC that utilizes a small bore nasal cannula to generate higher velocities of gas delivery than its counterparts using large bore HFNC. HVNI can accomplish a complete purge of extrathoracic dead space and may be able to provide ventilatory support in patients with acute hypercapnic respiratory failure in addition to oxygenation support .

This study is necessary because, even though studies were being conducted to determine both the optimal technique for HFNO delivery and the clinical setting in which it is most useful, the best strategy for weaning from HVNI remains unknown. It has also not been established at what point a patient should be considered stable enough to attempt to start withdrawing the HVNI

ELIGIBILITY:
Inclusion Criteria:

* This study will include Patients over 18 years receiving respiratory support through HVNI for acute hypoxemic respiratory failure
* Those eligible for weaning according to European Respiratory Society weaning criteria

Exclusion Criteria:

I. Extensive facial trauma or burn II. Refusal to participate. III. Usual long-term treatment with NIV for chronic disease IV. Tracheotomy or other upper airway disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Total weaning period (from the first time of being ready to wean till 48h after liberation of HVNI) | 3 days
  period taken for liberation from HVNI

SECONDARY OUTCOMES:
weaning outcome | 1 week
  failed or succeeded liberation
ICU stay | 1month
  period of ICU stay

IPD SHARING:
Plan to Share IPD: Undecided